CLINICAL TRIAL: NCT00259714
Title: Hemodynamic and Hormonal Responses to Dialysate Sodium Individualization in Hemodialysis Patients
Brief Title: Dialysate Sodium Individualization in Hemodialysis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol was not feasible - only 1 of 18 enrollees completed procedures.
Sponsor: Yale University (Other)
Collaborators: Satellite Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0509000646; 1034978.1.R06791..721688.02
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Hemodialysis Patients
Keywords: hypertension; hemodialysis; sodium; dialysate; hemodynamics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dialysate sodium (Active Comparator): In the control phase of the study, the prescribed dialysate sodium is 140 mEq/L
  Interventions: Drug: standard dialysate sodium
- dialysate sodium individualization (Experimental): .Dialysate sodium level prescribed matches the subject's average pre-dialysis serum sodium ("individualized").
  Interventions: Drug: dialysate sodium individualization

INTERVENTIONS:
Drug: dialysate sodium individualization — Dialysate sodium level prescribed matches the subject's average pre-dialysis serum sodium ("individualized").
  Arms: dialysate sodium individualization
Drug: standard dialysate sodium — The prescribed dialysate sodium is 140 mEq/L
  Arms: standard dialysate sodium

SUMMARY:
Salt and water excess is an essential mechanism of hypertension. This is particularly relevant to patients with end stage kidney disease (ESKD) on dialysis. We have demonstrated that individualization of the sodium concentration in the dialysate as to match the patient's own serum sodium concentration leads to less thirst, interdialytic weight gain, and better BP control in hypertensive patients. In this study we will evaluate the mechanisms underlying this response by measuring systemic hemodynamics, body volume spaces, and biochemical marker of volume status.

DETAILED DESCRIPTION:
Recent evidence from our group shows that individualization of the sodium concentration in the dialysate to match the patient's own serum sodium results in less thirst, less interdialytic weight gain, less HD-related symptoms, and better blood pressure control in hypertensive subjects. In this project we will evaluate the effect of dialysate sodium individualization on systemic hemodynamics, body volume compartments and biochemical markers of volume control in hypertensive hemodialysis patients. We will use a single-blind cross-over design with randomized blocks. After a 3-week baseline period where pre-HD serum sodium will be measured weekly to establish each patient's average serum sodium, subjects will be randomized to 3 weeks on standard dialysate sodium (140 mmol/L) or individualized dialysate sodium (same concentration as the average pre-HD serum sodium during the baseline period), then crossed over to the other for another 3 weeks after a 1-week washout period (dialysate Na 140 mmol/L). The remainder of the dialysis prescription, prescribed dry weight and vasoactive drugs will remain unchanged throughout the study. Clinical information, pre/intra/post-HD blood pressure and thirst scores will be measured weekly at the mid-week dialysis session. In addition, we will measure systemic hemodynamics (cardiac output and systemic vascular resistance), bioimpedance measurements of intracellular and extracellular volume, arterial stiffness (aortic augmentation index, aortic pulse wave velocity), interdialytic (44h) ambulatory BP monitoring, and plasma BNP, renin, aldosterone and norepinephrine at baseline and at the end of each block.

ELIGIBILITY:
Inclusion Criteria:

* ESKD on hemodialysis
* Hypertension, defined as average pre-HD BP >150/85 mmHg or use of antihypertensive drugs
* Average pre-HD serum sodium <139 mmol/L

Exclusion Criteria:

* Intradialytic hypotension
* Atrial fibrillation or other chronic tachyarrhythmia (due to effects on measuring equipment)
* Uncontrolled hypertension (average pre-HD BP >200/105 mmHg)
* Uncontrolled diabetes mellitus (due to problems on interpretation of serum sodium values)
* Debilitating illness
* Inability to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
BP changes on 44-h ABPM | 3 weeks
Changes in cardiac output and systemic vascular resistance | 3 weeks
Changes in intracellular and extracellular volume | 3 weeks

SECONDARY OUTCOMES:
Changes in measured biochemical markers | 3 weeks
Changes in augmentation index | 3 weeks
Change in circadian BP profile on 44-h ABPM | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aldo J Peixoto, MD, Principal Investigator — Yale University and VA Connecticut Healthcare System
Locations (1):
- Davita New Haven Dialysis Unit, New Haven, Connecticut, United States

REFERENCES:
- [Background] de Paula FM, Peixoto AJ, Pinto LV, Dorigo D, Patricio PJ, Santos SF. Clinical consequences of an individualized dialysate sodium prescription in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1232-8. doi: 10.1111/j.1523-1755.2004.00876.x. PMID 15327422